CLINICAL TRIAL: NCT04504682
Title: Neuraxial Analgesia With and Without Ambulation in Laboring Nulliparous Obese Women
Brief Title: Ambulation With Labor Epidural in Obese Women
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Limited recruitment
Sponsor: University of Chicago (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB19-1600
Record Dates: First submitted 2020-08-06; First posted 2020-08-07 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Obesity; Labor Onset and Length Abnormalities
MeSH Terms: conditions — Obesity | interventions — Walking

STUDY DESIGN:
Masking Description: The person completing analysis will be blinded to the treatment group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ambulation (Experimental): Participants in this arm will be encouraged to ambulate with epidural in place.
  Interventions: Behavioral: Ambulation

INTERVENTIONS:
Behavioral: Ambulation — Patients will be encouraged to ambulate for 20 minutes of every hour.

SUMMARY:
The purpose of this study is to determine if ambulation with a labor epidural in place is associated with decreased rate of cesarean delivery in obese patients.

DETAILED DESCRIPTION:
Obese women are known to have increased risk of cesarean delivery and prolonged labors. Low concentration epidural analgesia can achieve pain relief and allow for ambulation. Prior investigations have not shown a benefit in cesarean delivery between those who ambulate with an epidural and those who do not. These studies were conducted in women with normal weights. It is unknown if ambulation with a labor epidural is beneficial in decreasing cesarean delivery among obese women.

Obese women at term with a singleton pregnancy will be enrolled in this pilot study. Patients will receive their epidural analgesia when they desire per standard protocol at our institution. Following epidural placement, a Modified Bromage Score and straight leg test will be performed. If the patient passes the straight leg test and has a modified Bromage score > 6, they will be allowed to ambulate. They will be encouraged to ambulate for 20 minutes per hour with another adult alongside them. Obstetric care will be standard of care.

On postpartum day one, the patient will be administered a Labor Agentry Scale. Chart review will then be conducted to review maternal and neonatal outcomes.

ELIGIBILITY:
Inclusion Criteria:

Subjects capable of giving consent Singleton pregnancy Nulliparous (defined as no previous pregnancy beyond 20 weeks 0 days) Gestational age greater than or equal to 37 weeks BMI > = 35 at time of delivery admission Adult companion available Anticipated vaginal delivery

Exclusion Criteria:

Physical disability precluding ambulation Magnesium Administration Contraindications to neuraxial analgesia Cerclage in current pregnancy Active labor DPE Category III fetal heart tracing Fetal Demise In Utero

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2020-08-25 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

PRIMARY OUTCOMES:
Cesarean Delivery Rate | At time of delivery
  Percent of cesarean delivery

SECONDARY OUTCOMES:
Labor Duration | From labor onset to time of delivery
  Duration (hrs)
First Stage Duration | From onset of labor until complete dilation
  Duration (hrs)
Second Stage Duration | From complete dilation until delivery
  Duration (hrs)
Perceived Labor Control | Within 4 days postpartum
  Score on Labor Agentry Scale

CONTACTS AND LOCATIONS:
Overall Officials: Maritza Gonzalez, Principal Investigator — Faculty
Locations (1):
- University of Chicago, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vallejo MC, Firestone LL, Mandell GL, Jaime F, Makishima S, Ramanathan S. Effect of epidural analgesia with ambulation on labor duration. Anesthesiology. 2001 Oct;95(4):857-61. doi: 10.1097/00000542-200110000-00012. PMID 11605924
- [Background] Collis RE, Harding SA, Morgan BM. Effect of maternal ambulation on labour with low-dose combined spinal-epidural analgesia. Anaesthesia. 1999 Jun;54(6):535-9. doi: 10.1046/j.1365-2044.1999.00802.x. PMID 10403865
- [Background] Karraz MA. Ambulatory epidural anesthesia and the duration of labor. Int J Gynaecol Obstet. 2003 Feb;80(2):117-22. doi: 10.1016/s0020-7292(02)00339-9. PMID 12566183
- [Background] Vahratian A, Zhang J, Troendle JF, Savitz DA, Siega-Riz AM. Maternal prepregnancy overweight and obesity and the pattern of labor progression in term nulliparous women. Obstet Gynecol. 2004 Nov;104(5 Pt 1):943-51. doi: 10.1097/01.AOG.0000142713.53197.91. PMID 15516383
- [Background] Nuthalapaty FS, Rouse DJ, Owen J. The association of maternal weight with cesarean risk, labor duration, and cervical dilation rate during labor induction. Obstet Gynecol. 2004 Mar;103(3):452-6. doi: 10.1097/01.AOG.0000102706.84063.C7. PMID 14990405